CLINICAL TRIAL: NCT00391274
Title: Phase 3 Study of Pemetrexed Versus Docetaxel in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Who Have Had Prior Chemotherapy
Brief Title: Chemotherapy for Patients With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10717; H3E-MC-JMID (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Results first posted 2010-03-30 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed (Experimental)
  Interventions: Drug: pemetrexed
- Docetaxel (Active Comparator)
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m2, intravenous (IV) every 21 days until disease progression, death or 12 months after enrollment
  Other Names: LY231514; Alimta
  Arms: Pemetrexed
Drug: docetaxel — 75 mg/m2, intravenous (IV), every 21 days until disease progression, death or 12 months after enrollment
  Arms: Docetaxel

SUMMARY:
The purpose of this study is to compare the efficacy and toxicity of pemetrexed and docetaxel administered on a 3-weekly schedule in the treatment of patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) who have had prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis NSCLC (Stage IIIA, IIIB, or IV), not amenable to curative surgery or radiotherapy
* At least one prior chemotherapy for palliative therapy
* Response Evaluation Criteria In Solid Tumors (RECIST) criteria for disease status assessment
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2

Exclusion Criteria:

* Concurrent administration of any other tumor therapy
* Pregnant or breast feeding
* Serious concomitant disorders
* Inability or unwillingness to take folic acid or vitamin B12 supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- China (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tianjin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan

REFERENCES:
- [Derived] Wu YL, Sun Y, Zhou CC, Zhang L, Yu SY, Ma SL, Han LL, Zhang XQ, Orlando M. Survival without common toxicity criteria grade 3/4 toxicity following second-line treatment with pemetrexed for nonsquamous non-small cell lung cancer in Chinese patients. Chin Med J (Engl). 2013;126(24):4624-8. PMID 24342300
- [Derived] Sun Y, Wu YL, Zhou CC, Zhang L, Zhang L, Liu XY, Yu SY, Jiang GL, Li K, Qin SK, Ma SL, Han L, Quinlivan M, Orlando M, Zhang XQ. Second-line pemetrexed versus docetaxel in Chinese patients with locally advanced or metastatic non-small cell lung cancer: a randomized, open-label study. Lung Cancer. 2013 Feb;79(2):143-50. doi: 10.1016/j.lungcan.2012.10.015. Epub 2012 Nov 20. PMID 23182660
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed | Docetaxel
Started | 107 | 104
Received at Least One Dose of Study Drug | 106 | 102
Completed | 46 | 47
Not Completed | 61 | 57
Not completed — Death Due to Study Disease | 55 | 45
Not completed — Lost to Follow-up | 0 | 3
Not completed — Physician Decision | 4 | 2
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Death Due to Adverse Event | 1 | 3
Not completed — Death Due to Indeterminate Cause | 1 | 0
Not completed — Death Not Study Related | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed | Docetaxel | Total
Number analyzed (Participants) | 107 | 104 | 211
Age Continuous [Mean (Standard Deviation); unit: years] | 56.4 (9.33) | 55.9 (11.41) | 56.1 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 43 | 77
  Male | 73 | 61 | 134
Race/Ethnicity, Customized [Number; unit: participants]
  East Asian | 107 | 104 | 211
Region of Enrollment [Number; unit: participants]
  China | 107 | 104 | 211
Basis for Pathological Diagnosis [Number; unit: participants]
  Cytological | 34 | 35 | 69
  Histopathological | 73 | 69 | 142
Disease Stage [Number; unit: participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage IIIA - the cancer has spread to nearby tissue or spread to far away lymph nodes; Stage IIIB - cancer spread to opposite side of chest, more than one tumor within same lobe of lung; Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver.
  participants
    Stage IIIA | 2 | 2 | 4
    Stage IIIB | 24 | 18 | 42
    Stage IV | 81 | 84 | 165
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 11 | 16 | 27
    1 - Ambulatory, Restricted Strenuous Activity | 84 | 77 | 161
    2 - Ambulatory, No Work Activities | 12 | 11 | 23
Number of Sites of Metastatic Disease [Number; unit: participants]
  1 Site | 10 | 15 | 25
  2 Sites | 32 | 31 | 63
  3 Sites | 34 | 30 | 64
  4 Sites | 11 | 12 | 23
  5 Sites | 11 | 8 | 19
  6 Sites | 4 | 8 | 12
  7 Sites | 3 | 0 | 3
  8 Sites | 1 | 0 | 1
  9 Sites | 0 | 0 | 0
  10 Sites | 1 | 0 | 1
Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma | 75 | 73 | 148
  Carcinoma, Squamous Cell | 27 | 25 | 52
  Mixed Cell Carcinoma, Lung | 3 | 3 | 6
  Missing | 2 | 3 | 5
Smoking Status [Number; unit: participants]
  Never Smoked | 50 | 49 | 99
  Smoked, But Quit | 53 | 44 | 97
  Currently Smoking | 4 | 11 | 15

OUTCOME MEASURES:

1. Secondary Outcome: Overall Tumor Response
Description: Response based on Response Evaluation Criteria In Solid Tumors (RECIST), which define when cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments. CR (complete response) = disappearance of all target lesions; PR (partial response) = 30% decrease in the sum of the longest diameter of target lesions; PD (progressive disease) = 20% increase in the sum of the longest diameter of target lesions; SD (stable disease) = small changes that do not meet above criteria.
Time Frame: baseline to measured tumor response (up to 24 months after study enrollment)
Population: Patients who received at least one dose of study drug and qualified for tumor response analysis (met following criteria: histologic or cytologic diagnosis of NSCLC that was not amenable to curative therapy; no concurrent systemic chemotherapy; presence of measurable or evaluable disease).
Measure: Number; unit: participants
Arm/Group | Pemetrexed | Docetaxel
Number analyzed (Participants) | 104 | 98
participants
  Complete Response | 0 | 0
  Partial Response | 10 | 4
  Stable Disease | 33 | 46
  Progressive Disease | 49 | 36
  Early Death from Malignant Disease | 7 | 6
  Early Death from Other Causes | 1 | 1
  Unknown | 4 | 5
Statistical Analysis 1: Comparison: Pemetrexed vs Docetaxel; Test type: Superiority or Other; p = 0.1326, Regression, Logistic — Logistic regression of best overall tumor response (complete response + partial response); Treatment was the only covariate; Odds Ratio (OR) = 2.50, 95% CI [0.76 to 8.25]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) time was defined as the time from the date of study enrollment to the date of the first of the following events: objective disease progression or death due to any cause. For patients who were alive and had not progressed, PFS was censored at the last contact.
Time Frame: baseline to measured progressive disease (up to 24 months after study enrollment)
Population: Intent to treat population. Patient censored:
  pemetrexed=25, docetaxel=39.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed | Docetaxel
Number analyzed (Participants) | 107 | 104
months | 2.8 [1.8 to 3.1] | 3.1 [2.8 to 3.7]
Statistical Analysis 1: Comparison: Pemetrexed vs Docetaxel; Test type: Superiority or Other; p = 0.7704, Log Rank
Statistical Analysis 2: Comparison: Pemetrexed vs Docetaxel; Test type: Superiority or Other; p = 0.7784, Regression, Cox; Treatment was the only covariate; Hazard Ratio (HR) = 1.05, 95% CI [0.75 to 1.46]

3. Secondary Outcome: Duration of Response
Description: Duration of tumor response is the duration from date of first objective status assessment of a complete or partial response to the first date of progression or death from any cause. For each patient who is not known to have died or to have had a progression of disease as of the data inclusion cut-off date, duration of tumor response was censored at the time of last prior contact. Due to the low number of patients in the analysis, the median duration of tumor response could not be calculated for the docetaxel arm. Available data are presented as "Number of Patients with Disease Progression".
Time Frame: time of response to progressive disease (up to 24 months)
Population: Patients who qualified for response (met following criteria: histologic or cytologic diagnosis of NSCLC that was not amenable to curative therapy; no concurrent systemic chemotherapy; presence of measurable or evaluable disease). Results not presented because median was not calculable for the docetaxel arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed | Docetaxel
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pharmacology Toxicity
Description: Maximum common terminology criteria (CTC) Grade 3 or 4 toxicities possibly related to study drug are reported. The worst grade event per cycle is reported. Grades range from 0 (none) to 5 (death). Grade 3 events are severe and Grade 4 events are life-threatening.
Time Frame: first dose of study drug up to 24 months
Population: Patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed | Docetaxel
Number analyzed (Participants) | 106 | 102
participants
  Serum Glutamic Pyruvic Transaminase | 1 | 0
  Hemoglobin | 7 | 3
  Leukocytes | 4 | 21
  Lymphopenia | 1 | 0
  Neutrophils/Granulocytes | 5 | 29
  Platelets | 7 | 0
  Hypokalemia | 0 | 1
  Anorexia | 1 | 0
  Constipation | 0 | 1
  Diarrhea | 0 | 5
  Enteritis | 0 | 1
  Fatigue (Asthenia, Lethargy, Malaise) | 3 | 5
  Febrile Neutropenia | 2 | 4
  Infection (Clinical/Microbiological: Neutrophils) | 0 | 1
  Infection (Unknown: Pneumonia) | 0 | 1
  Mucositis/Stomatitis | 1 | 0
  Neuropathy: Motor | 0 | 1
  Pain: Thorax Not Otherwise Specified (NOS) | 0 | 1
  Pericardial Effusion (Non-Malignant) | 1 | 0
  Pulmonary/Upper Respiratory - Other | 1 | 0
  Rash/Desquamation | 1 | 0

5. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of study enrollment to the date of death due to any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up. An amendment allowed for the collection of overall survival on an additional 43 survival events. At the time the original record was released, it was not possible to provide results with the 95% Confidence Interval (CI) since the upper limit was not calculable. The median and 95% CIs are now reported.
Time Frame: baseline to date of death from any cause (up to 24 months after study enrollment); amendment (up to 30 months after study enrollment)
Population: Intent to treat population. Number of patients censored (up to 24 months): pemetrexed = 51, docetaxel = 55. Number of participants censored (up to 30 months): pemetrexed = 30, docetaxel = 32.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed | Docetaxel
Number analyzed (Participants) | 107 | 104
months
  Overall Survival (up to 24 months) | 11.7 [8.7 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 12.2 [9.1 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
  Overall Survival (up to 30 months) | 11.4 [8.6 to 13.4] | 11.5 [8.9 to 15.2]
Statistical Analysis 1: Comparison: Pemetrexed vs Docetaxel; Test type: Superiority or Other; p = 0.4921, Regression, Cox — P-value for Overall Survival (up to 24 months); Treatment was the only covariate; Hazard Ratio (HR) = 1.14, 95% CI [0.78 to 1.68]
Statistical Analysis 2: Comparison: Pemetrexed vs Docetaxel; Test type: Superiority or Other; p = 0.9256, Regression, Cox — P-value for Overall Survival (up to 30 months); Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.74 to 1.40]

6. Post Hoc Outcome: Number of Patients With Disease Progression
Description: Number of patients who have died or have had progression of disease. This outcome substitutes for the outcome on Duration of Response.
Time Frame: time of response to progressive disease (up to 12 months)
Population: Patients who qualified for response (met following criteria: histologic or cytologic diagnosis of NSCLC that was not amenable to curative therapy; no concurrent systemic chemotherapy; presence of measurable or evaluable disease). Patients censored: pemetrexed=6, docetaxel=3.
Measure: Number; unit: participants
Arm/Group | Pemetrexed | Docetaxel
Number analyzed (Participants) | 10 | 4
participants | 4 | 1

ADVERSE EVENTS:
Arm/Group | Pemetrexed | Docetaxel
Serious Adverse Events (participants affected / at risk) | 10/106 | 12/102
Other Adverse Events (participants affected / at risk) | 99/106 | 95/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=106) | Docetaxel (N=102)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Resulted in death in one pemetrexed patient.
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — Resulted in death in one docetaxel patient.
Fatigue (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Resulted in death in one docetaxel patient.
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) — Resulted in death in one docetaxel patient.
Shock (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=106) | Docetaxel (N=102)
Anaemia (Blood and lymphatic system disorders) | 9 (13) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Leukopenia (Blood and lymphatic system disorders) | 4 (6) | 6 (14)
Abdominal distension (Gastrointestinal disorders) | 6 (8) | 3 (3)
Constipation (Gastrointestinal disorders) | 8 (12) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 15 (20)
Nausea (Gastrointestinal disorders) | 21 (26) | 12 (14)
Vomiting (Gastrointestinal disorders) | 19 (23) | 5 (7)
Chest pain (General disorders) | 6 (6) | 11 (12)
Fatigue (General disorders) | 48 (70) | 42 (71)
Oedema peripheral (General disorders) | 3 (5) | 6 (11)
Pyrexia (General disorders) | 17 (25) | 15 (22)
Nasopharyngitis (Infections and infestations) | 6 (7) | 1 (1)
Pneumonia (Infections and infestations) | 8 (10) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 6 (6)
Alanine aminotransferase increased (Investigations) | 33 (55) | 10 (10)
Aspartate aminotransferase increased (Investigations) | 23 (32) | 6 (7)
Haemoglobin decreased (Investigations) | 19 (19) | 16 (17)
Neutrophil count decreased (Investigations) | 13 (20) | 30 (71)
Platelet count decreased (Investigations) | 8 (11) | 5 (6)
White blood cell count decreased (Investigations) | 15 (23) | 31 (91)
Anorexia (Metabolism and nutrition disorders) | 38 (54) | 30 (40)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (11) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4) | 8 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (34) | 24 (30)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (38) | 22 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 18 (18)
Rash (Skin and subcutaneous tissue disorders) | 21 (31) | 4 (4)

LIMITATIONS AND CAVEATS:
The primary outcome measure of this trial was designed to include pooled data. In addition, the results for the outcome on Duration of Response could not be presented due to the low number of patients being analyzed in the docetaxel group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days